CLINICAL TRIAL: NCT06850233
Title: The Validation of a Coronary Artery Disease Screening Algorithm Based on Facial Photos in Community Population
Brief Title: The Validation of a CAD Screening Algorithm Based on Facial Photos in Community Population
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-ZX050
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Artificial Intelligence
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Algorithm external validation group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a coronary heart disease screening algorithm based on facial photos in community population.

ELIGIBILITY:
Inclusion Criteria:

* Community population with a pre-test probability greater than 5% for coronary artery disease

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft (CABG)
* The history of heart failure
* With artificially facial alteration (i.e. cosmetic surgery, facial trauma or make-up)
* Other situations which make patients fail to be photographed

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the algorithm | at the end of enrollment (6 months)
  The sensitivity of the CAD screening algorithm assessed in the group
Specificity of the algorithm | at the end of enrollment (6 months)
  The specificity of the CAD screening algorithm assessed in the group

SECONDARY OUTCOMES:
Discriminative capabilities | at the end of enrollment (6 months)
  Area under receiver operating curve (AUC) of the algorithm assessed in the group
Positive predictive value (PPV) | at the end of enrollment (6 months)
  PPV of the CAD screening algorithm assessed in the group
Negative predictive value (NPV) | at the end of enrollment (6 months)
  NPV of the CAD screening algorithm assessed in the group
Diagnostic accuracy rate | at the end of enrollment (6 months)
  Diagnostic accuracy rate of the algorithm assessed in the group

CONTACTS AND LOCATIONS:
Locations (1):
- People's Road Community Health Service Center, Zhoukou, Henan, China